CLINICAL TRIAL: NCT00983996
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Alendronate Sodium Tablets (10 mg; Mylan) and Fosamax Tablets (10 mg; Merck) in Healthy Volunteers
Brief Title: Fasting Study of Alendronate Sodium Tablets (10 mg) and Fosamax Tablets (10 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ALEN-0243
Record Dates: First submitted 2009-09-21; First posted 2009-09-24 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alendronate Sodium Tablets, 10 mg
  Interventions: Drug: Alendronate Sodium Tablets, 10 mg
- 2 (Active Comparator): Fosamax Tablets, 10 mg
  Interventions: Drug: Fosamax Tablets, 10 mg

INTERVENTIONS:
Drug: Alendronate Sodium Tablets, 10 mg — 10 mg, single-dose fasting
  Arms: 1
Drug: Fosamax Tablets, 10 mg — 10 mg, single-dose fasting
  Arms: 2

SUMMARY:
The objective of this study is to investigate the bioequivalence of Mylan's alendronate sodium 10 mg tablets to Merck's Fosamax 10 mg tablets following a single, oral 40 mg (4 x 10 mg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy, adult subjects, 18 years and older
* able to swallow medication

Exclusion Criteria:

* institutionalized subjects
* history of any significant disease
* use of any prescription or OTC medications within 14 days of start of study
* received any investigational products within 30 days prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-06; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | urine collection up to 36 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Insitute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com